CLINICAL TRIAL: NCT02600299
Title: Effectiveness of a Psycho-educational Group (PEG) Intervention on Supportive Care and Survivorship Issues in Early-stage Breast Cancer Survivors Who Have Received Systemic Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Alexandre Chan, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201504-00102
Record Dates: First submitted 2015-11-04; First posted 2015-11-09 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer; Cancer; Anxiety; Cognitive Dysfunction
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Anxiety Disorders; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Arm (Experimental): On the basis of previous studies that evaluated PEG interventions for women with breast cancer, a structured program based on the Cognitive Behavioral Therapy (CBT) principles was developed. Patients in the PEG group will be involved in three sessions of psychoeducation. The PEG program is designed to cover the various aspects outlined by the IOM on quality cancer survivorship. This program is designed to take place on three individual days on a weekend. For each session, three major topics will be covered, with lectures and interactive workshop integrated. Sessions will be conducted by healthcare professionals who are experts/well-versed in their respective domains.
  Interventions: Behavioral: Psychoeducation group
- Usual Care (Placebo Comparator): No active intervention provided.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Psychoeducation group — On the basis of previous studies that evaluated PEG interventions for women with breast cancer, a structured program based on the Cognitive Behavioral Therapy (CBT) principles was developed. Patients in the PEG group will be involved in three sessions of psychoeducation. The PEG program is designed to cover the various aspects outlined by the IOM on quality cancer survivorship.
  Arms: Intervention Arm
Behavioral: Usual Care — Usual Care
  Arms: Usual Care

SUMMARY:
As cancer mortality rates improve in Asia, there is an increasing focus on patient-reported outcomes and survivorship issues. In view of the numerous medication and psychosocial issues that are commonly faced by early-stage breast cancer survivors, it deems important to develop and conduct specific interventional programs to mitigate these problems. In the literature, it is well recognized that psychosocial interventions are effective to manage emotional distress and quality of life, with the evidence clearly clustered in studies on female patients with breast cancer. One meta-analysis suggested that psycho-oncologic interventions including individual psychotherapy, group psychotherapy, psychoeducation, relaxing training can produce positive effects on emotional distress, anxiety and depression, and health-related QOL.

The investigators hypothesize that a significant reduction in anxiety, improvement of cognition and improvement of health-related quality of life among those who receive psycho-education, in comparison to those in the usual care. Hence, this randomized trial is designed to assess the effectiveness of a psycho-educational group (PEG) intervention on supportive care and survivorship issues, which include anxiety, depression, cognitive function, toxicities management of cancer- or treatment- related physical symptoms, and health-related quality of life in early-stage breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with breast cancer were included if they met the following criteria:

  * 21 years or older
  * able to read and understand either English or Mandarin
  * diagnosis of Stages 1-3 breast cancer by a medical oncologist
  * completed adjuvant cytotoxic treatment

Exclusion Criteria:

* Diagnosed with severe psychiatric diagnosis such as severe cognitive disorders, mood disorders (psychiatric disorders requiring hospitalization) or serious personality disorders).

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Severity of anxiety, as measured using Beck Anxiety Inventory | Within one month after the program
Quality of life | Within one month after the program

SECONDARY OUTCOMES:
Severity of cognitive dysfunction, as measured using FACT-Cog | Within one month after the program
Severity of symptom burden, as measured using Rotterdam Symptom Checklist | Within one month after the program

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Chan, PharmD, Principal Investigator — National University of Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Chan A, Gan YX, Oh SK, Ng T, Shwe M, Chan R, Ng R, Goh B, Tan YP, Fan G. A culturally adapted survivorship programme for Asian early stage breast cancer patients in Singapore: A randomized, controlled trial. Psychooncology. 2017 Oct;26(10):1654-1659. doi: 10.1002/pon.4357. Epub 2017 Jan 25. PMID 28024163